CLINICAL TRIAL: NCT06634303
Title: Hybernia Delta H (ΔH) Brain Cooling System for: Post-Mechanical Endovascular Cerebral Cooling
Brief Title: Hybernia Medical Post-Mechanical Thrombectomy Cerebral Cooling in Stroke
Acronym: Post-MECC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hybernia Medical (Industry)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HM001
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Ischemic Stroke; Brain cooling; Cerebral Hypothermia; Neuroprotection; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Fist-in-human investigational device study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Post-Mechanical Cerebral Cooling (Experimental): Acute ischemic stroke patients undergoing mechanical thrombectomy.
  Interventions: Device: Brain cooling

INTERVENTIONS:
Device: Brain cooling — Brain cooling intervention in acute ischemic stroke patients post mechanical thrombectomy

SUMMARY:
Reducing the temperature of tissue or organs (hypothermia) produces a protective state, through multiple molecular mechanisms, against adverse effects that arise from disrupted organ blood flow, e.g. in acute ischemic stroke (AIS). AIS is often caused by a blood clot that occludes a brain artery which, in turn disrupts brain blood flow. In large vessel occlusions, the current standard includes mechanical thrombectomy (MT), a minimally-invasive procedure that aims at removing the clot via endovascular means. In this case, brain cooling can lead to protection (neuroprotection) not only from the adverse effects of stroke/ischemia itself, but also from complications arising from sudden re-opening of the blocked artery through primary treatment, MT. This potential complication of MT is called reperfusion injury.

In this first-in-human investigational deivce study, Hybernia Medical's endovascular brain cooling system will be applied in acute ischemic stroke patients undergoing MT. Post-MT, selective brain hypothermia will be induced and maintained over 30 minutes. Endpoints of this study include, clinical safety, device performance/usability, and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 89
2. Informed signed consent obtained from patient or legally authorized representative
3. Clinical symptoms consistent with acute ischemic stroke
4. Pre-stroke modified Rankin Scale (mRS) score 0-1
5. National Institute of Health Stroke Scale (NIHSS) ≥ 6
6. Alberta Stroke Program Early CT Score (ASPECTS) score 5-10
7. IV tissue plasminogen activator (tPA) or Tenecteplase (TNK) may be administered within 4.5h of last known well (LKW), if patient eligible
8. Mechanical thrombectomy (MT) treatment performed with arterial puncture within 24h of LKW.
9. Pre-MT catheter angiogram shows target occlusion in intracranial ICA, M1 MCA, or M2 MCA
10. End of MT catheter angiogram shows achievement of moderate-to-complete reperfusion (modified Treatment in Cerebral Ischemia score or mTICI 2a-3)

Exclusion Criteria:

1. Pre-MT CT or MRI shows acute intracranial hemorrhage.
2. Previous intracranial hemorrhage, AVM, neoplasm (except small meningioma), or vascular stent-implant
3. Coma or reduced level of consciousness prior to MT (NIHSS 1A>1)
4. Seizure between LKW and time of potential enrollment
5. Severe contrast allergy or absolute contraindication to iodinated contrast.
6. Hypersensitivity to cold, i.e., history of cold-sensitive antibodies, Raynaud syndrome, or hepatitis C
7. Hematocrit <33%
8. Severe known renal impairment, i.e., requires renal replacement therapy (dialysis).
9. Post-reperfusion investigational therapy cannot be started within 150 min following pre-treatment CT or MR imaging
10. Presumed septic embolism, suspicion of bacterial endocarditis.
11. Known pregnancy (in women with child-bearing potential)
12. Body weight < 40kg
13. Patient not willing and able to participate in follow-up visits to day 90.
14. Life expectancy <6 months due to pre-existing conditions such as severe heart or renal failure, cancer, etc.
15. Currently or within past 30 days participating in another investigational treatment study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Device Feasibility | During the intervention
  Completion of Brain Cooling over 30 minutes

SECONDARY OUTCOMES:
Any Intracranial Hemorrhage | Up to 7 days after the intervention
  Any radiologic confirmed intracranial hemorrhage as detected on follow-up CT.
Symptomatic Intracranial Hemorrhage | Up to 7 days after the intervention
  Associated with NIHSS reduction of ≥4 points or death
Serious Adverse Events | Up to 7 days after the intervention
  Incidence of serious adverse device effect (SADE)
Hypothermia Effect on Vasculature | Up to 24 hours after the intervention
  Hypothermia effect on vasculature, such as vasospasm on cerebral angiogram or follow-up CTA
Mortality | Up to 3 months after the intervention
  Death
Hospital Readmission | Up to 3 months after the intervention
  Due to stroke
Device Performance and Usability | During the intervention
  * Device installation, setup, and use
  * Circuit performance
  * Cooling performance and accuracy
  * Correct trigger of alarms
Final modified Treatment in Cerebral Infarction (mTICI) score | Pre-intervention
  Grade 0: no perfusion
  Grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion
  Grade 2 Grade 2a: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory (e.g. in one major division of the middle cerebral artery (MCA) and its territory)
  Grade 2b: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory (e.g. in two major divisions of the MCA and their territories)
  Grade 2c: near complete perfusion except for slow flow or distal emboli in a few distal cortical vessels
  Grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches
Infarct Size | 3 days after the intervention and up to 7 days after the intervention
  Final infarct size/volume
Global Disability via modified Rankin Scale (mRS) | Month 1 and Month 3 after the intervention
  mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke.
  (0) No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

OTHER OUTCOMES:
Time to Reperfusion | Pre-intervention
  Time from Symptom onset-to-Groin puncture and Time from CT-to-Puncture
Reperfusion Time | Pre-intervention
  Time from Puncture-to-Reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ribo, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mangla S, Choi JH, Barone FC, Novotney C, Libien J, Lin E, Pile-Spellman J. Endovascular external carotid artery occlusion for brain selective targeting: a cerebrovascular swine model. BMC Res Notes. 2015 Dec 21;8:808. doi: 10.1186/s13104-015-1714-7. PMID 26689288
- [Background] Dumitrascu OM, Lamb J, Lyden PD. Still cooling after all these years: Meta-analysis of pre-clinical trials of therapeutic hypothermia for acute ischemic stroke. J Cereb Blood Flow Metab. 2016 Jul;36(7):1157-64. doi: 10.1177/0271678X16645112. Epub 2016 Apr 18. PMID 27089911
- [Background] Wu C, Zhao W, An H, Wu L, Chen J, Hussain M, Ding Y, Li C, Wei W, Duan J, Wang C, Yang Q, Wu D, Liu L, Ji X. Safety, feasibility, and potential efficacy of intraarterial selective cooling infusion for stroke patients treated with mechanical thrombectomy. J Cereb Blood Flow Metab. 2018 Dec;38(12):2251-2260. doi: 10.1177/0271678X18790139. Epub 2018 Jul 18. PMID 30019993
- [Background] Wan Y, Tian H, Wang H, Wang D, Jiang H, Fang Q. Selective intraarterial hypothermia combined with mechanical thrombectomy for acute cerebral infarction based on microcatheter technology: A single-center, randomized, single-blind controlled study. Front Neurol. 2023 Feb 16;14:1039816. doi: 10.3389/fneur.2023.1039816. eCollection 2023. PMID 36873429
- [Background] Neimark MA, Konstas AA, Lee L, Laine AF, Pile-Spellman J, Choi J. Brain temperature changes during selective cooling with endovascular intracarotid cold saline infusion: simulation using human data fitted with an integrated mathematical model. J Neurointerv Surg. 2013 Mar;5(2):165-71. doi: 10.1136/neurintsurg-2011-010150. Epub 2012 Jan 22. PMID 22270331
- [Background] Choi JH, Pile-Spellman J. Reperfusion Changes After Stroke and Practical Approaches for Neuroprotection. Neuroimaging Clin N Am. 2018 Nov;28(4):663-682. doi: 10.1016/j.nic.2018.06.008. PMID 30322601
- [Background] Choi JH, Pile-Spellman J. Selective brain hypothermia. Handb Clin Neurol. 2018;157:839-852. doi: 10.1016/B978-0-444-64074-1.00052-5. PMID 30459044
- [Background] Choi JH, Poli S, Chen M, Nguyen TN, Saver JL, Matouk C, Pile-Spellman J. Selective Brain Hypothermia in Acute Ischemic Stroke: Reperfusion Without Reperfusion Injury. Front Neurol. 2020 Nov 13;11:594289. doi: 10.3389/fneur.2020.594289. eCollection 2020. PMID 33281733
- [Background] Konstas AA, Neimark MA, Laine AF, Pile-Spellman J. A theoretical model of selective cooling using intracarotid cold saline infusion in the human brain. J Appl Physiol (1985). 2007 Apr;102(4):1329-40. doi: 10.1152/japplphysiol.00805.2006. Epub 2006 Dec 14. PMID 17170208
- [Background] Choi JH, Marshall RS, Neimark MA, Konstas AA, Lin E, Chiang YT, Mast H, Rundek T, Mohr JP, Pile-Spellman J. Selective brain cooling with endovascular intracarotid infusion of cold saline: a pilot feasibility study. AJNR Am J Neuroradiol. 2010 May;31(5):928-34. doi: 10.3174/ajnr.A1961. Epub 2010 Jan 6. PMID 20053807